CLINICAL TRIAL: NCT04514757
Title: Transcutaneous (Tragus) Vagal Nerve Stimulation (tVNS) for Post-op Atrial Fibrillation (POAF)
Brief Title: Transcutaneous (Tragus) Vagal Nerve Stimulation for Post-op Afib
Acronym: STOP_AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Jonathan K. Ho, Associate Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-001636
Record Dates: First submitted 2020-07-29; First posted 2020-08-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: post-operative atrial fibrillation; transcutaneous (tragus) vagal nerve stimulation; outcomes
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Active tVNS (Parasym device, Parasym Health, Inc, London, UK) will be performed with a clip attached to ear at 20 Hz, 250ms at a current just below discomfort threshold for one hour twice a day, starting on post-day 0. Stimulation will continue until 5 days post-operatively or discharge.
  Interventions: Device: active tVNS
- Control Group (Sham Comparator): Sham tVNS will be performed by attaching the Parasym device to the ear and setting output to 0. Stimulation will continue until 5 days post-operatively or discharge.
  Interventions: Device: sham tVNS

INTERVENTIONS:
Device: active tVNS — 20 Hz, 250ms at a current just below discomfort threshold for one hour twice a day, starting on post-day 0. Stimulation will continue until 5 days post-operatively or discharge.
  Arms: Intervention Group
Device: sham tVNS — Current set a 0 mA, starting on post-op day 0. Stimulation will continue until 5 days post-operatively or discharge.
  Arms: Control Group

SUMMARY:
Patients undergoing cardiac surgery are at high risk of developing atrial fibrillation (AF), with estimated rates of 30-50% and occurs at approximately 2-4 days after surgery. The autonomic nervous system is known to play a key role in AF. Animal studies have indicated that duration and inducibility of AF can be decreased with intermittent vagus nerve stimulation (VNS). In humans, literature suggests that transcutaneous (tragus) VNS (tVNS) can serve as a potentially non-invasive therapy for treatment of post-operative AF (POAF) by reducing inflammation and increasing atrial refractory period. The purpose of this study is to determine the value of tVNS in reducing the burden of POAF and days of hospitalization after cardiac surgery.

DETAILED DESCRIPTION:
The trial will have two study arms: active tVNS vs. sham tVNS. Patients will be randomized to active tVNS vs. sham tVNS and will receive optimal post-op care in both arms. Active tVNS (Parasym device, Parasym Health, Inc, London, UK) will be performed with a clip attached to the ear at 20 hertz (Hz), 250 microseconds (ms) at a current just below discomfort threshold for one hour twice a day, starting on post-day 0. For sham tVNS, Parasym device will be attached to the ear twice a day, turned on but current set to 0 milliamp (mA), starting on post-op day 0. Stimulation will continue until 5 days post-op or discharge. Discomfort threshold will be determined in both arms pre-operatively in the conscious state. This current will be used for stimulation for this patient until they are awake and extubated after surgery. The stimulation threshold may be reassessed once the patient is able to provide feedback.

Patients will be approached and recruited prior to their scheduled cardiac surgery. Recruited patients who give informed consent will have the discomfort stimulation threshold (current that leads to discomfort at the tragus) determined prior to surgery. Post-operatively, stimulation will be performed in the tVNS group at just below discomfort threshold. In the sham group, the stimulator will be turned on but current set at 0 mA. Stimulations will be performed within 12 hours of arrival to the ICU after surgery, and then twice a day between the hours of 7:00-9:00 am and 6:00-8:00 pm. If POAF develops in either arm, stimulation will be continued for the full 5 days. Ten ml of blood will be drawn within 12 hours of arrival to the ICU after surgery and on day 3 post-op for measurement of biomarkers. Serum will be stored at -80 Celsius and processed in batches of 10-15 samples.

Sample Size:

The investigators expect cardiac surgery to be associated with 40% incidence of POAF. The investigators expect tVNS to reduce this incidence by 40%. A sample size of 133 subjects per arm will be able to achieve 80% power at alpha of 0.05. If interim analysis is planned, Pocock method will be used and a p value of 0.03 will be used for interim and 0.03 for final analysis. Data will be analyzed according to the intention-to-treat principle.

Randomization:

A 1:1 randomization ratio for the tVNS vs. sham will be utilized. Patients who meet all of the inclusion and none of the exclusion criteria will be randomized in the order of their enrollment. After completing the Informed Consent process, the subject is then randomized following completion of the baseline and demographics information case report forms. Randomization should occur prior to any study-related tests or procedures. The subjects will be considered enrolled in the study once randomization has occurred.

Randomization will be stratified by clinical center and post-operative amiodarone use. A computer-generated randomization list with random permuted block of a variable will be produced for each clinical center. Investigators and other study staff members should not be able to identify the study assignment until this time. If a randomization assignment is inadvertently disclosed prior to use, the assignment will never be used.

A report of randomization compliance will be generated at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo coronary artery bypass surgery, major vascular/aneurysm repair requiring bypass, valvular replacement or repair, or both, for clinically indicated reasons.
2. Age ≥ 18 years.
3. Sinus rhythm at baseline.
4. Provision of signed informed consent and stated willingness to comply with all study procedures for duration of the study

Exclusion Criteria:

1. Emergent surgery
2. Anticipated amiodarone use
3. Patients with permanent or persistent atrial fibrillation
4. Planned concomitant atrial Maze procedure
5. Complex congenital heart disease
6. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal).
7. Left ventricular assist device or status post orthotopic heart or lung transplantation
8. Unable or unwilling to comply with protocol requirements.
9. Known channelopathy such as Brugada syndrome, long QT syndrome, or Catecholaminergic monomorphic ventricular tachycardia
10. Symptomatic sinus bradycardia or sinus node dysfunction at baseline without an implantable pacemaker.
11. Complete heart block or trifascicular block without an implantable pacemaker
12. Recurrent vasovagal syncope
13. Unilateral or bilateral vagotomy
14. Chronic amiodarone use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation | 6 days
  Incidence of post-operative atrial fibrillation for postoperative day 0-5 (postop day 0 is the day of the surgery and is the first day of the time frame and postoperative day 5 is the 6th day).

SECONDARY OUTCOMES:
Days of hospitalization | Postop day 0 until discharge from the hospital, an average of 1 week.
  Number of days in the hospital from postoperative day 0 to discharge.
Inflammatory markers | Within 12 hours of arrival to the ICU after surgery and on postop day 3 (2 days)
  Reduction in inflammatory markers including C-reactive protein (CRP), Interleukin 10 (IL-10), Tumour Necrosis Factor alpha (TNF-alpha), Interleukin 6 (IL-6), and Interleukin 1 beta (IL-1β)
Sympathetic neural markers | Postop day 3 (1 day)
  Reduction in sympathetic neural markers including norepinephrine, Neuropeptide Y (NPY), and galanin.
Pain assessment | 6 days
  Pain scores will be assessed on postoperative days 0-5 using the visual analog score (Scale 0-10). Zero for no pain and ten being the worst pain experienced. They will be obtained and recorded into the medical record by the nurse monitoring the subject as part of standard care. Postop day 0 is the day of the surgery and is the first day of the time frame and postoperative day 5 is the 6th day.
Narcotic Usage | 6 days
  Total narcotic consumption will be calculated each day for postoperative days 0-5. Narcotic amount will be converted to a standard unit equivalent for comparison. Postop day 0 is the day of the surgery and is the first day of the time frame and postoperative day 5 is the 6th day.
Duration of post-op atrial fibrillation | 6 days
  How many hours or days for each incidence of postoperative atrial fibrillation for postoperative days 0-5 (postop day 0 is the day of the surgery and is the first day of the time frame and postoperative day 5 is the 6th day).
Heart rate during atrial fibrillation | 6 days
  The heart rate during each incidence of postoperative atrial fibrillation for postop days 0-5 (postop day 0 is the day of the surgery and is the first day of the time frame and postoperative day 5 is the 6th day).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ho, MD, Principal Investigator — University of California, Los Angeles; Marmar Vaseghi, MD, Principal Investigator — University of California, Los Angeles; Stavros Stavrakis, MD, PhD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maisel WH, Rawn JD, Stevenson WG. Atrial fibrillation after cardiac surgery. Ann Intern Med. 2001 Dec 18;135(12):1061-73. doi: 10.7326/0003-4819-135-12-200112180-00010. PMID 11747385
- [Background] Aranki SF, Shaw DP, Adams DH, Rizzo RJ, Couper GS, VanderVliet M, Collins JJ Jr, Cohn LH, Burstin HR. Predictors of atrial fibrillation after coronary artery surgery. Current trends and impact on hospital resources. Circulation. 1996 Aug 1;94(3):390-7. doi: 10.1161/01.cir.94.3.390. PMID 8759081
- [Background] Chen PS, Chen LS, Fishbein MC, Lin SF, Nattel S. Role of the autonomic nervous system in atrial fibrillation: pathophysiology and therapy. Circ Res. 2014 Apr 25;114(9):1500-15. doi: 10.1161/CIRCRESAHA.114.303772. PMID 24763467
- [Background] Salavatian S, Beaumont E, Longpre JP, Armour JA, Vinet A, Jacquemet V, Shivkumar K, Ardell JL. Vagal stimulation targets select populations of intrinsic cardiac neurons to control neurally induced atrial fibrillation. Am J Physiol Heart Circ Physiol. 2016 Nov 1;311(5):H1311-H1320. doi: 10.1152/ajpheart.00443.2016. Epub 2016 Sep 2. PMID 27591222
- [Background] Stavrakis S, Humphrey MB, Scherlag B, Iftikhar O, Parwani P, Abbas M, Filiberti A, Fleming C, Hu Y, Garabelli P, McUnu A, Peyton M, Po SS. Low-Level Vagus Nerve Stimulation Suppresses Post-Operative Atrial Fibrillation and Inflammation: A Randomized Study. JACC Clin Electrophysiol. 2017 Sep;3(9):929-938. doi: 10.1016/j.jacep.2017.02.019. Epub 2017 May 30. PMID 29759717
- [Background] Stavrakis S, Humphrey MB, Scherlag BJ, Hu Y, Jackman WM, Nakagawa H, Lockwood D, Lazzara R, Po SS. Low-level transcutaneous electrical vagus nerve stimulation suppresses atrial fibrillation. J Am Coll Cardiol. 2015 Mar 10;65(9):867-75. doi: 10.1016/j.jacc.2014.12.026. PMID 25744003
- [Background] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678
- [Background] Andreas M, Arzl P, Mitterbauer A, Ballarini NM, Kainz FM, Kocher A, Laufer G, Wolzt M. Electrical Stimulation of the Greater Auricular Nerve to Reduce Postoperative Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2019 Oct;12(10):e007711. doi: 10.1161/CIRCEP.119.007711. Epub 2019 Oct 10. PMID 31597476